CLINICAL TRIAL: NCT03808649
Title: Individualized Volume of Oral Contrast Agent Based on the Clinical Risk Factor in CT Enterography: a Randomized Controlled Trial
Brief Title: Individualized Volume of Oral Contrast Agent in CT Enterography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019SDU-QILU-01
Record Dates: First submitted 2019-01-12; First posted 2019-01-17 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: CTE
MeSH Terms: interventions — Mannitol

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized group (Active Comparator): Participants are given different volume of a preparation of mannitol based on BMI as oral contrast agent over an hour prior to the examination.
  Interventions: Drug: 1500ml of 2.5% mannitol; Drug: different volume of 2.5% mannitol
- conventional group (Experimental): Participants are given 1500ml of a preparation of mannitol as oral contrast agent over an hour prior to the examination.
  Interventions: Drug: 1500ml of 2.5% mannitol

INTERVENTIONS:
Drug: 1500ml of 2.5% mannitol — 1500ml of 2.5% mannitol was used in experimental group
Drug: different volume of 2.5% mannitol — different volume of 2.5% mannitol based on BMI was used in active comparator group
  Arms: Individualized group

SUMMARY:
Small bowel distension is mandatory for the assessment of the bowel wall in CT enterography, but some patients were sufferring inadequate small bowel distension. So, it is important to prescribe personalized regimen according to patient's personal characteristics.

DETAILED DESCRIPTION:
CT enterography has become an important tool in the evaluation of small bowel diseases, especially in patients with inflammatory bowel diseases. Small bowel distension is mandatory for the assessment of the bowel wall. So, it is important to find clinical risk factors for inadequate small bowel distension and prescribe personalized regimen according to patient's personal characteristics to reduce patient acceptance.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing CT enterography

Exclusion Criteria:

* patients with a history of GI surgery
* patients with known or suspected bowel obstruction or perforation
* patients with severe chronic renal failure (creatinine clearance<30 ml/min)
* patients with uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* patients with acute upper GI bleeding
* patients with severe inflammatory bowel disease or megacolon
* patients with documented allergy to intravascular contrast agent
* patients with pregnancy or lactation
* patients hemodynamically unstable
* patients unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-01-20 (Estimated); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-07-20 (Estimated)

PRIMARY OUTCOMES:
Clinical risk factors for inadequate small bowel distention | 2 month
  Number of clinical risk factors for inadequate small bowel distention
Adequate small bowel distention | 4 month
  The assessment system includes four parts
  1. Whether the contrast reached the caecum is evaluate and recorded as "yes" or "no"
  2. The overall presence of inhomogeneous contrast is evaluated and recorded as "yes" or "no"
  3. The maximum dimension of a single loop in each quadrant was recorded.
  4. The scale of loops of small bowel distended are evaluated and recorded as "0%-25%","26%-50%","51%-75%","75%-100%"

SECONDARY OUTCOMES:
Side effects | 4 month
  Side effects in 2 groups The degree of nausea, emesis, diarrhea, abdominal distension and cramp following ingestion are scored on a scale ranging from 0 to 4, in which a higher score represents a higher level of these targets.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China